CLINICAL TRIAL: NCT04305145
Title: Phase II Study of Infliximab for the Treatment of Immune Checkpoint Inhibitor Colitis
Brief Title: Infliximab for Treatment of Immune Checkpoint Inhibitor Colitis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Michael Dougan, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19-763
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Melanoma Stage III; Melanoma Stage IV; Skin Cancer Stage III; Skin Cancer Stage IV; Drug-Induced Colitis; Drug Toxicity; Immune-related Adverse Event
Keywords: Melanoma; Skin cancer; Drug toxicity; Colitis; Immune checkpoint inhibitor; Immunotherapy toxicity; Immune-related adverse event
MeSH Terms: conditions — Melanoma; Skin Neoplasms; Drug-Related Side Effects and Adverse Reactions; Colitis | interventions — Infliximab; Methylprednisolone; Methylprednisolone Hemisuccinate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Infliximab (Experimental): Patients randomized to this arm will receive IV infliximab regardless of whether they are hospitalized due to their colitis.
  * Infliximab: Predetermined dose of intravenous infliximab, up to 3 times over 7 weeks
  * Crossover for inadequate response: Patients who do not respond to initial treatment within 3 days with a decrease in symptoms by one grade, or who do not improve to grade 2 or less symptoms by 5 days will add combination therapy from the other treatment arm (corticosteroids) at full initial dosing.
  Interventions: Drug: Infliximab
- Corticosteroids (Experimental): Patients randomized to this arm will receive IV steroids or oral steroids depending on whether the severity of their colitis requires hospitalization ("inpatient").
  * Inpatient: Predetermined intravenous dose of methylprednisolone, 2x daily up until patients can safely be transitioned to an oral prednisone taper
  * Outpatient: Predetermined oral dose of predisone, daily over 7 weeks
  Crossover for inadequate response: Patients who do not respond to initial treatment within 3 days with a decrease in symptoms by one grade, or who do not improve to grade 2 or less symptoms by 5 days will add combination therapy from the other treatment arm (infliximab) at full initial dosing.
  Interventions: Drug: Methylprednisolone; Drug: Prednisone

INTERVENTIONS:
Drug: Infliximab — Infusion
  Other Names: AVSOLA; Ixifi; Remicade; Renflexis
  Arms: Infliximab
Drug: Methylprednisolone — Infusion
  Other Names: Solu-Medrol; Duralone; Medralone; Medrol; M-Prednisol
  Arms: Corticosteroids
Drug: Prednisone — Orally
  Other Names: Deltasone; Prednicot; predniSONE Intensol; Rayos; Sterapred; Sterapred DS
  Arms: Corticosteroids

SUMMARY:
The goal of this clinical trial is to compare the safety and effectiveness of infliximab compared to steroids for the treatment of immune checkpoint inhibitor-induced colitis (ICI colitis) in patients with stage III/IV skin cancer.

The main questions this study aims to answer are:

* How many patients treated with infliximab experience steroid-free disease resolution after 7 weeks?
* How many patients treated with steroids experience steroid-free disease resolution after 7 weeks?

DETAILED DESCRIPTION:
This is a phase II, randomized, signal-detection trial to evaluate the efficacy and safety of the drugs infliximab, methylprednisolone, and prednisone to manage the side of effect of colitis caused by immune checkpoint inhibitors (ICIs) that target a protein called CTLA-4. An example of one of these ICIs is ipilimumab, which has been approved by the FDA to treat metastatic melanoma.

The names of the treatments involved in this study are:

* Infliximab
* Methylprednisolone
* Prednisone

The FDA has approved infliximab, methylprednisolone, and prednisone to treat many conditions affecting the immune system, including colitis.

Participants will receive a CTLA-4 inhibitor, like ipilimumab, and any other cancer treatments as part of their regular care for stage III/IV skin cancer at the discretion of treating oncologist.

Participants who enroll in this study will undergo one or more flexible sigmoidoscopies or colonoscopies as part of their clinical care. The first of these procedures would occur at the time of study enrollment, and the second may occur after several weeks of treatment at the discretion of the study doctor. During these procedures, biopsies will be collected for clinical purposes as well as for research purposes. Blood will also be collected for research at the time of enrollment and at the time of study completion. Any extra samples for research would only be collected if it is safe for the participant.

Participants will also complete weekly follow-ups either over the phone or in-person that may last about 10 minutes. During these visits, participants will be asked about any new symptoms or changes in their health, their medications, and their GI symptoms. Blood for research may be collected at one or more of these visits if it coincides with a scheduled clinical blood draw.

Participants are expected to be on study treatment for approximately 7 weeks. Once participants complete the study treatment, the study team will review their medical records every 6 months for any changes in their health.

It is expected that about 42 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Stage III/IV skin cancer
* Treatment with CTLA-4 inhibitor alone or in combination with PD-1or PD-L1 blockade within the past 8 weeks
* Clinically significant diarrhea resulting in the decision to pause immunotherapy treatment
* Endoscopically visible colitis (Mayo 1-3) at the time of screening

Exclusion Criteria:

* Prior history of inflammatory colitis related to immune checkpoint inhibitors requiring treatment with > 10 mg/day of prednisone or equivalent, or any other immunosuppressive medication
* Concurrent immune-related Adverse Event (irAE) requiring treatment with systemic corticosteroids (dose equivalent of prednisone 10 mg/day or higher) or another systemic immune suppressing medication within the past 10 days
* Current use of any immune suppressing biologic medication, or use within the last 4 weeks; immune stimulating medications such as checkpoint blockade are explicitly permitted
* Current use of combination treatment with an investigation immunotherapy targeting a pathway other than PD-1 or PD-L1, concurrent chemotherapy, or targeted therapy
* Previous adverse reaction to infliximab or corticosteroids
* Colonic perforation or abscess present at the time of screening
* History of Hepatitis B or C with a positive viral load, untreated mycobacterium tuberculosis, or active herpes zoster infection
* Current bacterial infection requiring antibiotic treatment, or systemic fungal infection
* Prior history of inflammatory bowel disease, microscopic colitis or segmental colitis associated with diverticulosis
* Received more than 3 doses of systemic corticosteroids, or receive dsystemic corticosteroids at a dose exceeding 2mg/kg methylprednisolone or equivalent, within 72 hours prior to endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-08-31 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with Steroid-Free Colitis | 7 weeks
  Proportion of Patients with Steroid-Free Colitis at seven weeks with steroid-free colitis remission defined as less than 7.5 mg a day of prednisone or equivalent and grade-1 or lower symptoms.

SECONDARY OUTCOMES:
Proportion of Participants with Treatment Related Adverse Events as Assessed by CTCAE 5. | 6 Months
  National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
The proportion of patients requiring secondary immune suppression-Infliximab | 7 Weeks
  patients randomly assigned to infliximab, secondary immune support will be defined as requiring subsequent treatment with steroids. The proportions of patients in each treatment arm requiring secondary immune suppression will be summarized and presented with 90% exact binomial confidence intervals
The proportion of patients requiring secondary immune suppression-Steroids | 7 Weeks
  patients randomly assigned to steroids, secondary immune support will be defined as requiring subsequent treatment with steroids. The proportions of patients in each treatment arm requiring secondary immune suppression will be summarized and presented with 90% exact binomial confidence intervals
Time to steroid-free remission | randomization to grade-1 or lower symptoms of colitis and less than 7.5 mg a day of prednisone or equivalent or up to 6 months
  The initial analysis of steroid-free remission will be based on cumulative incidence (1-Kaplan-Meier estimates).
Rate of Symptom Remission at 72 hours | 72 hours
  The proportion of patients in each treatment arm who have colitis symptom reduction to grade-1 or less within 72 hours of starting randomized treatment will be summarized and presented with 90% exact binomial confidence intervals. The treatment arms will be compared using Fisher's exact tests.
Rate of Symptom Remission at 4 Weeks | 4 weeks
  The proportion of patients in each treatment arm who have colitis symptom reduction to grade-1 or less within 72 hours of starting randomized treatment will be summarized and presented with 90% exact binomial confidence intervals. The treatment arms will be compared using Fisher's exact tests.
Proportion of patients with colectomy or colitis-specific mortality | 7 weeks
  The proportions of patients with colectomy or colitis-specific mortality (investigator assessed) will be presented by treatment arm with 90% exact binomial confidence intervals
Cumulative steroid exposure | 7 weeks
  Cumulative steroid exposure over time for each patient will be calculated by adding the number of doses multiplied by strength of dose over the total follow-up time. Steroid exposure will be summarized descriptively for each treatment arm, and compared using a Wilcoxon rank-sum test.
  With 20 patients per treatment arm, a Wilcoxon rank-sum test will have 80% power to detect a 41difference in cumulative steroid exposure that is 0.85 times the common standard deviation, assuming a one-sided, type-I error of 10
Progression Free Survival | duration of time from start of randomization to time of progression or death, whichever occurs first or up to 24 months.
  summarized using the method of Kaplan-Meier and compared using stratified log-rank tests
Overall Survival | the duration of time from start of randomization to time of death or up to 24 months
  summarized using the method of Kaplan-Meier and compared using stratified log-rank tests
Overall Response Rate | proportion of evaluable patients who achieve either a (complete response) CR or (partial response) PR or up to 24 Months
  Response rates will be summarized by treatment arm and presented with 90% exact binomial confidence intervals. The comparison of response rates between treatment arms will use Fisher's exact test

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dougan, MD, PHD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Massachusetts General Hospital (MGH) - Contact the Partners Innovations team at http://www.partners.org/innovation